CLINICAL TRIAL: NCT06210451
Title: Lubricant Gel Versus Sterile Water for Speculum Insertion During Embryo Transfer: a Randomized Non-inferiority Clinical Trial
Brief Title: Speculum Insertion During Embryo Transfer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Yossi Mizrachi, Principal Investigator, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0147-23-WOMC
Record Dates: First submitted 2023-12-18; First posted 2024-01-18 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: IVF
Keywords: IVF; Embryo transfer; Gel; RCT

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gel group (Experimental): Speculum insertion using sterile water-based gel
  Interventions: Other: Sterile water-based gel
- Sterile water group (No Intervention): Speculum insertion using sterile water

INTERVENTIONS:
Other: Sterile water-based gel — Insertion of the speculum during ET will be performed using 5 gr of water-based, sterile gel
  Arms: Gel group

SUMMARY:
Lubrication gels are widely used in numerous gynecologic procedures in order to ease the insertion of speculum and visualize the cervix. It was shown that applying lubricating gels significantly decreases patient pain during vaginal speculum examination. While many fertility specialists use lubrication gels to insert the speculum during embryo transfer (ET), others are strongly reluctant to use gels due to concern that they might have a detrimental effect on embryos and ET success. Similar concern was prevalent regarding the use of lubrication gel during Pap-smear for detection of cervical dysplasia. However, several studies have shown that the use of small amount of water-soluble gel does not change cervical cytology. Lubrication gels might have deleterious effect on sperm motility. However, there wasn't any study examining the effect of lubricant gel on ET success.

The investigators hypothesize that using a lubrication gel will not reduce the live birth rate per transfer, but decrease patient pain during procedure.

DETAILED DESCRIPTION:
In vitro fertilization (IVF) involves a highly complex series of events leading to the creation of an embryo. The transfer of that embryo, the final step in the process, is seen as a critical moment at the culmination of this incredibly intricate process. The technique of the embryo transfer (ET) has undergone a slow evolution, but for many physicians, this step remains relatively consistent throughout years of practice. While the procedure itself is relatively short, physicians often have specific preferences for each of the steps involved, either supported by evidence, learned from mentors or guided by experience and individual success. As such, ET success rates are a statistic that generates significant pride among physicians and are often tracked by clinics as a quality control metric. Interestingly, there are significant outcome differences between physicians.

Numerous techniques and practices employed during ET have been studied. For some, the evidence is robust, while for others, it is very limited. Some practices and techniques were found to improve ET success, such as: abdominal US guidance, removal of cervical mucus, use of a soft catheter, and placement of the embryo at a distance of more than 10 mm from the uterine fundus. For other aspects of ET there is no sufficient evidence to decide on the preferred practice. These include the optimal length of the procedure and rotation of the catheter during withdrawal. Good-quality randomized clinical trials are much needed in order to decide on the best practice. For example, there was previously a concern that the use of powdered gloves during ET might be toxic to the embryos. However, a single RCT (n=712) has shown that using powdered gloves resulted in similar pregnancy rates compared to unpowdered gloves.

Lubrication gels are widely used in numerous gynecologic procedures in order to ease the insertion of speculum and visualize the cervix. It was shown that applying lubricating gels significantly decreases patient pain during vaginal speculum examination. While many fertility specialists use lubrication gels to insert the speculum during ET, others are strongly reluctant to use gels due to concern that they might have a detrimental effect on embryos and ET success. Similar concern was prevalent regarding the use of lubrication gel during Pap-smear for detection of cervical dysplasia. However, several studies have shown that the use of small amount of water-soluble gel does not change cervical cytology. Lubrication gels might have deleterious effect on sperm motility. However, there wasn't any study examining the effect of lubricant gel on ET success.

The investigators hypothesize that using a lubrication gel will not reduce the live birth rate per transfer, but decrease patient pain during procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40
* Fresh and thawed ET
* Patients undergoing their 1st-3rd ET
* ET of 1-2 embryos

Exclusion Criteria:

* Age>40
* Egg donation cycles

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 416 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy or live birth rate. | 3 years
  Number of patients with ongoing pregnancy or live birth at >20 week's gestation.

SECONDARY OUTCOMES:
Positive serum BHCG | 3 years
  Number of patients with positive serum BHCG test.
Clinical pregnancy | 3 years
  Number of patients with transvaginal ultrasound test demonstrating fetal cardiac activity.
Questionnaire | 3 years
  Pain score on a scale of 1 to 10, where 1 indicates no pain and 10 indicates worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Tairy, MD, Principal Investigator — Edith Wolfson Medical Center
Locations (1):
- Faculty of Medical and Health Sciences, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Yes
anonymous IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 years